CLINICAL TRIAL: NCT05808218
Title: WASH for Everyone: Testing Alternative Approaches to Sanitation and Hygiene Behaviour Change in Chiradzulu, Malawi
Acronym: W4E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Malawi University of Business and Applied Sciences (MUBAS) WASHTED Centre (Unknown); University of Strathclyde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 28249
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-10

CONDITIONS: Behavior
Keywords: sanitation; handwashing; hygiene
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CLTS (Experimental): This arm will receive a standard community-led total sanitation) intervention).
  Interventions: Other: Community-Led Total Sanitation
- CLTS Plus (Experimental): Includes all activities in the CLTS arm with the addition of village-level Care Groups for sanitation and hygiene promotion.
  Interventions: Other: Community-Led Total Sanitation; Other: Care Groups
- Control (No Intervention)

INTERVENTIONS:
Other: Community-Led Total Sanitation — The community-led total sanitation intervention is implemented across an entire Traditional Authority and includes the following village-level activities:
  1. Triggering:
     * Village transect walks and open defecation site mapping
     * Demonstrations of food contamination and medical expense calculations
  2. Development of a Community-Action Plan and identification of "natural leaders"
  3. Post-triggering: routine follow-up by selected natural leaders to track and monitor progress against the Community Action Plan
  In addition to the activities above, the WASH for Everyone team will:
  * Train a cadre of local masons on sanitation construction
  * Support the District Health office in the implementation of existing sanitation and hygiene promotion at village markets and other public spaces
  Other Names: CLTS
  Arms: CLTS; CLTS Plus
Other: Care Groups — * Orientation and training of village-level Care Group members on CLTS, latrine construction, and hygiene promotion
  * Routine house-to-house follow-up of Care Group members to provide peer-to-peer counselling and support on sanitation and hygiene behaviours.
  Arms: CLTS Plus

SUMMARY:
This study aims to assess the impact of multiple community-based behaviour change approaches on sanitation and hygiene behaviours in rural Malawi. Three different sub-districts (Traditional Authorities) in Chiradzulu District will be selected, each receiving a different combination of community-based interventions or will serve as controls. Eligible communities, households, and individuals will be randomly selected in each Traditional Authority and sanitation and hygiene behaviours assessed through self-report and direct observation after 1 year of intervention.

DETAILED DESCRIPTION:
This is a controlled before-and-after study that will evaluate the impact on sanitation and hygiene behaviours of different community-based interventions implemented as part of the WASH For Everyone programme. WASH for Everyone, implemented by World Vision and Water For People. WASH for Everyone is a 3-year project (2022 - 2024) that aims to achieve universal access to water, sanitation, and hygiene (WASH) in Chiradzulu district, and promote improved sanitation and hygiene behaviours. There are two primary community-based sanitation and hygiene behaviour change approaches included in the WASH for Everyone interventions: 1) community-led total sanitation (CLTS), a widely implemented participatory approach to ending open defecation at the community-level and 2) Care Groups, a model using locally-based volunteer groups to implement peer-to-peer counselling and support with a long history in nutrition programming.

For the purposes of this study, one Traditional Authority will receive the CLTS intervention. A second Traditional Authority will receive the CLTS intervention with the additional of village-level Care Groups (CLTS +). A third traditional authority will serve as the comparison group.

Within study Traditional Authorities, communities will be selected at random for inclusion in the study. Twenty communities will be enrolled in both the CLTS and the CLTS+ Traditional Authorities. Thirty communities will be enrolled from the comparison Traditional Authority. In each selected community, an average of 20 households will be enrolled at baseline and again at endline. Difference-in-difference analysis will be used to measure the changes in primary and secondary outcomes between either intervention and control and between the two intervention groups.

ELIGIBILITY:
Households are primary sampling unit. Household eligibility requirements are:

Inclusion Criteria:

* Presence of an adult head of household age 18 or over who gives consent for the household to participate in the study; household is permanent resident of selected village

Exclusion Criteria:

* No permanent resident aged 18 or over; temporary resident of community/households

In selected households, 1 individual will be selected at random to complete study survey. Individual eligibility requirements are:

Inclusion criteria:

* Permanent resident of selected household; able to provide informed consent

Exclusion criteria:

* Not a permanent resident of selected household, not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2800 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
sanitation coverage | study endline (one year)
  Sanitation coverage is defined as confirmed presence of a functional sanitation facility in the home or compound that meets standard definitions of at least unimproved sanitation facilities according to the Joint Monitoring Programme. This will be determined by reported access to a private, household sanitation facility that respondents self-identify as completed. Self-reported access will be verified through visual inspection of the sanitation facilities.

SECONDARY OUTCOMES:
sanitation use | study endline (one year)
  Self-reported exclusive use of a sanitation facility for defecation among all members of a select households
safe disposal of child feces | study endline (one year)
  Self-reported disposal of feces of any child under the age of five in a latrine / toilet
handwashing facility | study endline (one year)
  presence of a dedicated device / location in the household were both soap and water are available for handwashing
Basic sanitation coverage | study endline (one year)
  coverage: basic sanitation coverage is defined as the presence of a completed sanitation facility at the home that meets the minimum criteria of a basic sanitation facility, i.e. improved facility not shared with other households
Sanitation-related Quality-of-Life Index | study endline (one year)
  Sanitation-related Quality of Life (SANQOL) is a five-question instrument for measuring the degree of achievement of the following sanitation-related capabilities: privacy, safety, health, shame and disgust. Scores range from 0 to 1 with higher scores indicating a higher sanitation-related quality of life.
Handwashing behaviour | study endline (one year)
  observed handwashing with soap at critical moments (after defecation, cleaning a child and before cooking, eating, or feeding a child); measured through a three-hour direct observation in 50% of all study participants

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dreibelbis, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Malawi University of Business and Applied Sciences, WASHTED Centre, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
All data will be fully anonymised and posted on a public repository for third party use. To completely anonymise the data prior to uploading it onto an open data site, any references to specific places, information about occupation, and any other information that holds the potential to identify the respondents will be redacted. Public repository will be determined in collaboration with study partners and project funders.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be made available within 1 year of final data collection

REFERENCES:
- [Derived] Chidziwisano K, Panulo M, MacLeod C, Vigneri M, White B, Wells J, Ross I, Morse T, Dreibelbis R. Water, Sanitation, and Hygiene for Everyone Intervention Study: Protocol for a Controlled Before-and-After Trial. JMIR Res Protoc. 2025 May 15;14:e68280. doi: 10.2196/68280. PMID 40373302